CLINICAL TRIAL: NCT05084781
Title: Arthroscopic Rotator Cuff Repair Utilizing Mechanical Bone Debridement Versus Coblation Debridement: A Prospective Randomized Double Blind Controlled Trial
Brief Title: Arthroscopic Rotator Cuff Repair Utilizing Mechanical Bone Debridement Versus Coblation Debridement
Acronym: FLOW90
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB19-1158
Record Dates: First submitted 2021-10-06; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: Paralle study arms for 1)coblation debridement, 2) mechanical debridement
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind - patient and outcome assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Coblation Debridement (Experimental): FLOW 90 / WEREWOLF debridement of rotator cuff footprint.
  Interventions: Procedure: Coblation Debridement (FLOW90)
- Mechanical Debridement (Active Comparator): Standard mechanical debridement of rotator cuff footprint.
  Interventions: Procedure: Coblation Debridement (FLOW90)

INTERVENTIONS:
Procedure: Coblation Debridement (FLOW90) — bipolar radiofrequency energy

SUMMARY:
Randomized controlled trial comparing coblation debridement to mechanical debridement in rotator cuff repair.

DETAILED DESCRIPTION:
Prospective, Double blind, Randomized controlled trial. Male and female subjects, over the age of 18 years. Full thickness rotator cuff tear, requiring surgical repair. Patient undergoes pre- and intra-operative assessment, and once eligibility is confirmed intra-operatively, patient is randomly assigned to receive either a) coblation debridment, or b) mechanical debridement.

Standard post-operative rehab program for all patients. Follow-up occurs at 3, 6, 12, and 24 months post operatively and includes physical exam and patient based outcomes (questionnaires).

ELIGIBILITY:
Inclusion Criteria:

1. The subject has signed the REB approved informed consent form (ICF) specific to this study prior to enrollment
2. The subject has a repairable full thickness rotator cuff tear with an estimated full thickness size <5cm confirmed with diagnostic MRI in AP or ML dimension and /or ultrasound
3. The subject is independent, ambulatory, and can comply with all post-operative evaluations and visits
4. The subject has persistent pain and functional disability and has failed conservative treatment (e.g. PT, steroid injection, anti-inflammatory) for > 3 months
5. The subject is at least eighteen (18) years of age and considered to be skeletally mature

Exclusion Criteria:

1. The subject has undergone previous rotator cuff repair surgery to the affected shoulder
2. The subject has a partial thickness rotator cuff tear
3. The subject requires a concomitant labral repair
4. The subject has an irreparable rotator cuff tear
5. The subject is unable or unwilling to undergo MRI scan.
6. The investigator judges the subject unlikely to remain compliant to follow-up.
7. The subject has received an investigational therapy or approved therapy for investigational use within 30 days prior to the surgery
8. The subject is a prisoner, or is known or suspected to be transient
9. The subject's condition represents a worker's compensation case
10. The subject is currently involved in a health-related litigation procedure
11. The subject currently has an acute infection in the area surrounding the surgical site
12. The subject has a major medical illness (life expectancy less than 2 years or unacceptably high operative risk
13. Fatty atrophy >50% (Goutallier grade 4-5)

INTRA-OPERATIVE EXCLUSIONS:

1. Massive or irreparable rotator cuff tear which cannot be mobilized to the midpoint of the footprint of the rotator cuff on the greater tuberosity
2. Co-existing labral pathology requiring repair with sutures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Western Ontario Rotator Cuff Score (WORC) | 24 months
  Shoulder based quality of life measurement tool

SECONDARY OUTCOMES:
Western Ontario Rotator Cuff Score (WORC) | 3 months, 6 months, 12 months
  Shoulder based quality of life measurement tool
Quick Disability of the Arm Shoulder and Hand (QuickDASH) questionnaire | 3 months, 6 months, 12 months, 24 months
  Short version of the DASH questionnaire for musculoskeletal disorders of the upper extremity
Re-tear of rotator cuff | 12 months
  Evaluated via MRI

CONTACTS AND LOCATIONS:
Overall Officials: Ian Lo, MD FRSCS, Principal Investigator — University of Calgary
Locations (1):
- Access Orthopaedics, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No